CLINICAL TRIAL: NCT01426763
Title: An Open-label Multiple-dose Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Subcutaneous Administration of CINRYZE® (C1 Esterase Inhibitor [Human]) With Recombinant Human Hyaluronidase (rHuPH20) in Subjects With Hereditary Angioedema
Brief Title: A Study to Evaluate the Safety and Pharmacology of Subcutaneous Administration of CINRYZE With Recombinant Human Hyaluronidase
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Collaborators: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0624-204; SPD616-204 (Other: Sponsor)
Record Dates: First submitted 2011-08-25; First posted 2011-08-31 (Estimated); Results first posted 2013-01-04 (Estimated); Last update posted 2021-07-19 (Actual); Status verified 2021-06

CONDITIONS: Hereditary Angioedema
Keywords: HAE; C1 esterase inhibitor; C1 INH; Subcutaneous; hyaluronidase; rHuPH20
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — SERPING1 protein, human; Complement C1 Inhibitor Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SC CINRYZE with rHuPH20 Dose Level 1 (Experimental): Subcutaneous injection of 1000 Units of CINRYZE with 20,000 Units of rHuPH20 twice weekly for two weeks
  Interventions: Biological: CINRYZE with rHuPH20
- SC CINRYZE with rHuPH20 Dose Level 2 (Experimental): Subcutaneous injection of 2000 Units of CINRYZE with 40,000 Units of rHuPH20 twice weekly for two weeks
  Interventions: Biological: CINRYZE with rHuPH20

INTERVENTIONS:
Biological: CINRYZE with rHuPH20
  Other Names: C1 esterase inhibitor (human); Recombinant human hyaluronidase

SUMMARY:
The objectives of the study are to:

1. Evaluate the safety and tolerability of subcutaneously administered CINRYZE with recombinant human hyaluronidase (rHuPH20) in subjects with hereditary angioedema (HAE) who previously participated in CINRYZE Study 0624-200 (NCT01095497)
2. Characterize the pharmacokinetics and pharmacodynamics of subcutaneously administered CINRYZE with rHuPH20
3. Assess the immunogenicity of CINRYZE following subcutaneous (SC) administration of CINRYZE with rHuPH20

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this protocol, a subject must:

1. Provide informed consent/assent, as appropriate.
2. Have previously participated in CINRYZE Study 0624-200 and completed the subcutaneous therapy period in that study.
3. During the 3 consecutive months prior to screening, have a history of less than 1 HAE attack per month (average) that required treatment with C1 INH therapy or other blood products.
4. Agree to avoid his/her known HAE triggers during the study to the best of his/her ability.

Exclusion Criteria:

To be eligible for this protocol, a subject must not:

1. Have received C1 INH therapy or any blood products for treatment or prevention of an HAE attack within 14 days prior to the first dose of study drug.
2. Have received any ecallantide (Kalbitor), icatibant (Firazyr), or antifibrinolytics (e.g., tranexamic acid) within 14 days prior to the first dose of study drug.
3. Have any change (start, stop, or change in dose) in androgen therapy (e.g., danazol, oxandrolone, stanozolol, testosterone) within 14 days prior to the first dose of study drug.
4. If female, have started taking or changed the dose of any hormonal contraceptive regimen or hormone replacement therapy (i.e., estrogen/progestin containing products) within 3 months prior to the first dose of study drug.
5. Have a history of abnormal blood clotting.
6. Have a history of allergic reaction to products containing C1 INH or other blood products.
7. Have a known allergy to hyaluronidase or any other ingredient in rHuPH20.
8. Be pregnant or breastfeeding.
9. Have received an investigational study drug within 30 days prior to the first dose of study drug.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-09-12 (Actual); Primary Completion 2011-11-28 (Actual); Study Completion 2011-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (4):
- United States (4):
  - ViroPharma Investigational Site, Scottsdale, Arizona
  - ViroPharma Investigational Site, Walnut Creek, California
  - ViroPharma Investigational Site, Atlanta, Georgia
  - ViroPharma Investigational Site, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Subcutaneous (SC) CINRYZE With Recombinant Human Hyaluronidase ph20 (rHuPH20) Dose Level 1: SC injection of 1000 Units of CINRYZE with ~20,000 Units of rHuPH20 twice weekly for two weeks
- SC CINRYZE With rHuPH20 Dose Level 2: SC injection of 2000 Units of CINRYZE with ~40,000 Units of rHuPH20 twice weekly for two weeks
Period: Overall Study
Arm/Group | Subcutaneous (SC) CINRYZE With Recombinant Human Hyaluronidase ph20 (rHuPH20) Dose Level 1 | SC CINRYZE With rHuPH20 Dose Level 2
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subcutaneous (SC) CINRYZE With Recombinant Human Hyaluronidase ph20 (rHuPH20) Dose Level 1 | SC CINRYZE With rHuPH20 Dose Level 2 | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (7.79) | 33.7 (10.27) | 32.6 (8.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Adverse Events, Number of Participants With Local Injection Site Reactions, and Number of Participants Who Discontinue Study Drug or Withdraw From the Study
Time Frame: 18 days
Measure: Number; unit: participants
Arm/Group | Subcutaneous (SC) CINRYZE With Recombinant Human Hyaluronidase ph20 (rHuPH20) Dose Level 1 | SC CINRYZE With rHuPH20 Dose Level 2
Number analyzed (Participants) | 6 | 6
participants
  Number of participants with adverse events | 6 | 5
  Number of participants with injection site reactions | 6 | 5
  Number of participants who discontinued study drug | 0 | 0
  Number of participants who withdrew from the study | 0 | 0

2. Secondary Outcome: Mean Change C1 Inhibitor (C1INH)
Description: Mean Change in Baseline in Observed Plasma Concentration of C1 Inhibitor (C1INH) Antigen. Baseline-corrected concentrations were derived by subtracting the observed pre-dose concentrations on Day 1 of each treatment period from each observed concentration.
Time Frame: 18 days
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: g/L
Groups:
- Subcutaneous (SC) With Recombinant Human Hyaluronidase ph20 (rHuPH20) CYNRYZE Dose 1: 1000 Units of SC CYNRYZE with ~20,000 Units of rHuPH20 twice weekly for two weeks
Arm/Group | Subcutaneous (SC) With Recombinant Human Hyaluronidase ph20 (rHuPH20) CYNRYZE Dose 1 | SC CINRYZE With rHuPH20 Dose Level 2
Number analyzed (Participants) | 6 | 6
g/L
  0 Hour (h) | 0.0248 (0.0565) | 0.00483 (0.00904)
  1 hour (h) post Dose 1 | 0.0273 (0.065) | 0.00383 (0.00417)
  2 h post Dose 1 | 0.0302 (0.0637) | 0.008 (0.0123)
  3 h post Dose 1 | 0.0275 (0.0602) | 0.0095 (0.00729)
  4 h post Dose 1 | 0.0382 (0.0652) | 0.011 (0.00537)
  6 h post Dose 1 | 0.0398 (0.0599) | 0.020 (0.00678)
  8 h post Dose 1 | 0.0455 (0.0624) | 0.031 (0.0154)
  24 h post Dose 1 | 0.0625 (0.0728) | 0.0612 (0.0212)
  48 h post Dose 1 | 0.0665 (0.0749) | 0.0603 (0.0213)
  Pre-Dose 2 | 0.0243 (0.0234) | 0.0507 (0.0168)
  1 h post Dose 2 | 0.0387 (0.0749) | 0.00833 (0.00852)
  120 h post Dose 1 | 0.020 (0.00883) | 0.0388 (0.0132)
  Pre-Dose 3 | 0.0288 (0.0644) | 0.00833 (0.0095)
  1 h post Dose 3 | 0.00217 (0.00271) | 0.004 (0.00405)
  Pre-Dose 4 | 0.006 (0.0119) | 0.0128 (0.00854)
  1 h post Dose 4 | 0.0193 (0.012) | 0.033 (0.0196)
  2 h post Dose 4 | 0.0233 (0.0126) | 0.0377 (0.021)
  3 h post Dose 4 | 0.0238 (0.012) | 0.0333 (0.0163)
  4 h post Dose 4 | 0.0257 (0.0142) | 0.037 (0.0215)
  6 h post Dose 4 | 0.0298 (0.0124) | 0.039 (0.025)
  8 h post Dose 4 | 0.0354 (0.0118) | 0.0397 (0.0157)
  24 h post Dose 4 | 0.0347 (0.018) | 0.0623 (0.0207)
  48 h post Dose 4 | 0.0273 (0.0171) | 0.0562 (0.00906)
  72 h post Dose 4 | 0.0167 (0.0185) | 0.046 (0.0106)
  120 h post Dose 4 | 0.0165 (0.0214) | 0.0157 (0.00797)
  168 h post Dose 4 | 0.00933 (0.0201) | 0.0382 (0.0935)

3. Secondary Outcome: Mean Change C4 Compliment
Description: Mean Change in Baseline in Observed Plasma Concentration of C4 Compliment. Baseline-corrected concentrations were derived by subtracting the observed pre-dose concentrations on Day 1 of each treatment period from each observed concentration.
Time Frame: 18 days
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Subcutaneous (SC) With Recombinant Human Hyaluronidase ph20 (rHuPH20) CYNRYZE Dose 1 | SC CINRYZE With rHuPH20 Dose Level 2
Number analyzed (Participants) | 6 | 6
mg/L
  0 Hour (h) | 9.00 (15.4) | 13.3 (14.4)
  1 hour (h) post Dose 1 | 11.0 (14.3) | 10.3 (21.4)
  2 h post Dose 1 | 11.3 (13.8) | 11.0 (18.7)
  3 h post Dose 1 | 10.2 (11.7) | 11.5 (17.6)
  4 h post Dose 1 | 11.5 (13.6) | 13.2 (16.8)
  6 h post Dose 1 | 15.7 (14.2) | 14.0 (18.1)
  8 h post Dose 1 | 16.3 (16.6) | 22.5 (29.1)
  24 h post Dose 1 | 25.0 (15.6) | 30.5 (19.5)
  48 h post Dose 1 | 37.4 (23.1) | 49.8 (24.3)
  Pre-Dose 2 | 24.3 (14.5) | 53.3 (23.2)
  1 h post Dose 2 | 37.5 (21.6) | 53.2 (22.6)
  120 h post Dose 1 | 35.6 (22.6) | 70.8 (28.4)
  Pre-Dose 3 | 29.0 (19.1) | 66.3 (47.0)
  1 h post Dose 3 | 32.5 (18.7) | 69.3 (50.5)
  Pre-Dose 4 | 32.0 (18.4) | 62.5 (54.2)
  1 h post Dose 4 | 30.2 (18.8) | 57.3 (53.7)
  2 h post Dose 4 | 33.3 (24.5) | 59.7 (52.5)
  3 h post Dose 4 | 34.3 (17.9) | 53.3 (46.2)
  4 h post Dose 4 | 34.8 (22.9) | 63.3 (56.5)
  6 h post Dose 4 | 36.3 (21.6) | 59.7 (46.4)
  8 h post Dose 4 | 33.6 (20.3) | 56.5 (48.4)
  24 h post Dose 4 | 37.8 (23.0) | 64.7 (52.4)
  48 h post Dose 4 | 33.0 (22.4) | 65.7 (47.0)
  72 h post Dose 4 | 23.3 (20.6) | 72.2 (57.5)
  120 h post Dose 4 | 16.8 (15.5) | 58.7 (46.4)
  168 h post Dose 4 | 19.0 (18.4) | 44.8 (46.0)

4. Secondary Outcome: Number of Subjects With C1 INH Antibodies
Time Frame: Day 1 (pre-dose), Day 18 (168 h post Dose 4), and 30 (±2) days after the last dose of study drug (Dose 4)
Measure: Number; unit: Participants
Groups:
- Subcutaneous (SC) With Recombinant Human Hyaluronidase ph20 (rHuPH20) CYNRYZE Dose 1: SC injection of 1000 Units of CINRYZE with ~20,000 Units of rHuPH20 twice weekly for two weeks
Arm/Group | Subcutaneous (SC) With Recombinant Human Hyaluronidase ph20 (rHuPH20) CYNRYZE Dose 1 | SC CINRYZE With rHuPH20 Dose Level 2
Number analyzed (Participants) | 6 | 6
Participants
  Day 1 (pre-dose) | 0 | 0
  Day 18 (168 h post Dose 4) | 0 | 0
  30 (±2) days after the last dose of study drug (Dose 4) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Subcutaneous (SC) CINRYZE With Recombinant Human Hyaluronidase ph20 (rHuPH20) Dose Level 1 | SC CINRYZE With rHuPH20 Dose Level 2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Subcutaneous (SC) CINRYZE With Recombinant Human Hyaluronidase ph20 (rHuPH20) Dose Level 1 (N=6) | SC CINRYZE With rHuPH20 Dose Level 2 (N=6)
Injection site erythema (General disorders) | 5 | 5 — Two subjects (one at each dose level) each reported two events of severe injection site erythema; all other adverse events reported in the study were of mild or moderate intensity.
Injection site hemorrhage (General disorders) | 1 | 0
Injection site induration (General disorders) | 0 | 1
Injection site edema (General disorders) | 1 | 0
Injection site pain (General disorders) | 4 | 1
Injection site pruritus (General disorders) | 1 | 0
Injection site swelling (General disorders) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement. Most restrictive provision - PI will not publish results until after first of: multicenter publication is published or 24 months from study end. Thereafter, PI may publish his results. PI must provide copy of proposed publication to Sponsor for pre-review. If Sponsor requests, PI must delete Sponsor confidential information before publication and/or delay publication for 60 days so Sponsor can file for patents or take other action to protect its patent rights.